CLINICAL TRIAL: NCT05348603
Title: Leveraging Community Engagement and Electronic Health Record Strategies to Promote Diverse Participation in Clinical Research
Brief Title: Electronic Health Record Strategies to Promote Diverse Participation in Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 2000032716; 75F40120C00174 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2022-04-19; First posted 2022-04-27 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Patient Participation
Keywords: Online Patient Portal
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: To examine the effectiveness of enhanced online patient portal features in increasing interest and participation in clinical trials, a randomized trial that will employ a full 2X2X2X2 factorial design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- No Intervention (No Intervention): *No intervention.
- Traditional Letter Only (Experimental): *A mailed letter will invite the patient to set up a research profile in their patient portal.
  Interventions: Other: Traditional Letter
- Direct to Patient Message Only (Experimental): *An e-mail sent to the patient will inform the patient that there is a message pending in their patient portal regarding opportunities to participate in research.
  Interventions: Other: Direct to Patient Message
- Chatbot Only (Experimental): *A real-time, interactive chatbot on the patient portal will encourage research participation and direct patients to learn more about research opportunities and trials that match their interests.
  Interventions: Other: Chatbot
- Banner Only (Experimental): *Banner-type "advertisements" will appear during routine viewing and use of of the patient's portal for their our medical/clinical care inform patients of research opportunities.
  Interventions: Other: Banner
- Traditional Letter + Direct to Patient Message (Experimental): * A mailed letter will invite the patient to set up a research profile in their patient portal; AND
  * An e-mail sent to the patient will inform the patient that there is a message pending in their patient portal regarding opportunities to participate in research.
  Interventions: Other: Traditional Letter; Other: Direct to Patient Message
- Traditional Letter + Chatbot (Experimental): * A mailed letter will invite the patient to set up a research profile in their patient portal; AND
  * A real-time, interactive chatbot will encourage research participation and direct patients to learn more about research opportunities and trials that match their interests.
  Interventions: Other: Traditional Letter; Other: Chatbot
- Traditional Letter + Banner (Experimental): * A mailed letter will invite the patient to set up a research profile in their patient portal; AND
  * Banner-type "advertisements" during routine viewing and use of of the patient's portal for their our medical/clinical care inform patients of research opportunities.
  Interventions: Other: Traditional Letter; Other: Banner
- Direct to Patient Message + Chatbot (Experimental): * An e-mail sent to the patient will inform the patient that there is a message pending in their patient portal regarding opportunities to participate in research; AND
  * A real-time, interactive chatbot will encourage research participation and direct patients to learn more about research opportunities and trials that match their interests.
  Interventions: Other: Direct to Patient Message; Other: Chatbot
- Direct to Patient Message + Banner (Experimental): * An e-mail sent to the patient will inform the patient that there is a message pending in their patient portal regarding opportunities to participate in research AND
  * Banner-type "advertisements" during routine viewing and use of of the patient's portal for their our medical/clinical care inform patients of research opportunities.
  Interventions: Other: Direct to Patient Message; Other: Banner
- Chatbot + Banner (Experimental): * A real-time, interactive chatbot will encourage research participation and direct patients to learn more about clinical trial opportunities and trials that match their interests; AND
  * Banner-type "advertisements" during routine viewing and use of of the patient's portal for their our medical/clinical care will inform patients of research opportunities.
  Interventions: Other: Chatbot; Other: Banner
- Traditional Letter + Direct to Patient Message + Chatbot (Experimental): * A mailed letter will invite the patient to set up a research profile in their patient portal; AND
  * An e-mail sent to the patient will inform the patient that there is a message pending in their patient portal regarding opportunities to participate in research; AND
  * A real-time, interactive chatbot will encourage research participation and direct patients to learn more about research opportunities and trials that match their interests.
  Interventions: Other: Traditional Letter; Other: Direct to Patient Message; Other: Chatbot
- Traditional Letter + Direct to Patient Message + Banner (Experimental): * A mailed letter will invite the patient to set up a research profile in their patient portal; AND
  * An e-mail sent to the patient will inform the patient that there is a message pending in their patient portal regarding opportunities to participate in research; AND
  * Banner-type "advertisements" during routine viewing and use of of the patient's portal for their our medical/clinical care inform patients of research opportunities.
  Interventions: Other: Traditional Letter; Other: Direct to Patient Message; Other: Banner
- Traditional Letter + Chatbot + Banner (Experimental): * A mailed letter will invite the patient to set up a research profile in their patient portal; AND
  * A real-time, interactive chatbot will encourage research participation and direct patients to learn more about research opportunities and trials that match their interests.
  AND
  *Banner-type "advertisements" during routine viewing and use of of the patient's portal for their our medical/clinical care inform patients of research opportunities.
  Interventions: Other: Traditional Letter; Other: Chatbot; Other: Banner
- Direct to Patient Message + Chatbot + Banner (Experimental): * An e-mail sent to the patient will inform the patient that there is a message pending in their patient portal regarding opportunities to participate in research; AND
  * A real-time, interactive chatbot will encourage research participation and direct patients to learn more about research opportunities and trials that match their interests; AND
  * Banner-type "advertisements" during routine viewing and use of of the patient's portal for their our medical/clinical care inform patients of research opportunities.
  Interventions: Other: Direct to Patient Message; Other: Chatbot; Other: Banner
- Traditional Letter + Direct to Patient Message + Chatbot + Banner (Experimental): * A mailed letter will invite the patient to set up a research profile in their patient portal; AND
  * An e-mail sent to the patient will inform the patient that there is a message pending in their patient portal regarding opportunities to participate in research; AND
  * A real-time, interactive chatbot will encourage research participation and direct patients to learn more about research opportunities and trials that match their interests; AND
  * Banner-type "advertisements" during routine viewing and use of of the patient's portal for their our medical/clinical care inform patients of research opportunities.
  Interventions: Other: Traditional Letter; Other: Direct to Patient Message; Other: Chatbot; Other: Banner

INTERVENTIONS:
Other: Traditional Letter — Patients receive a traditional letter.
  Arms: Traditional Letter + Banner; Traditional Letter + Chatbot; Traditional Letter + Chatbot + Banner; Traditional Letter + Direct to Patient Message; Traditional Letter + Direct to Patient Message + Banner; Traditional Letter + Direct to Patient Message + Chatbot; Traditional Letter + Direct to Patient Message + Chatbot + Banner; Traditional Letter Only
Other: Direct to Patient Message — Patients receive a direct to patient message via the portal.
  Arms: Direct to Patient Message + Banner; Direct to Patient Message + Chatbot; Direct to Patient Message + Chatbot + Banner; Direct to Patient Message Only; Traditional Letter + Direct to Patient Message; Traditional Letter + Direct to Patient Message + Banner; Traditional Letter + Direct to Patient Message + Chatbot; Traditional Letter + Direct to Patient Message + Chatbot + Banner
Other: Chatbot — Patients are contacted by a chatbot via the portal.
  Arms: Chatbot + Banner; Chatbot Only; Direct to Patient Message + Chatbot; Direct to Patient Message + Chatbot + Banner; Traditional Letter + Chatbot; Traditional Letter + Chatbot + Banner; Traditional Letter + Direct to Patient Message + Chatbot; Traditional Letter + Direct to Patient Message + Chatbot + Banner
Other: Banner — Patients are exposed to a banner ad via the portal.
  Arms: Banner Only; Chatbot + Banner; Direct to Patient Message + Banner; Direct to Patient Message + Chatbot + Banner; Traditional Letter + Banner; Traditional Letter + Chatbot + Banner; Traditional Letter + Direct to Patient Message + Banner; Traditional Letter + Direct to Patient Message + Chatbot + Banner

SUMMARY:
The purpose of this study is to determine the effectiveness of enhanced features in an online patient portal including banners, a chatbot, and direct to patient message and traditional mailed letters on increasing interest in research among online patient portal users.

DETAILED DESCRIPTION:
The primary objective is to examine the effectiveness of enhanced online patient portal features including banners, a chatbot, and direct to patient message and traditional mailed letters on increasing interest in research among online patient portal users, as measured by the user's creation of a research profile.

The secondary objective is to examine the effectiveness of two enhanced online patient portal features including banners, a chatbot and direct-to-patient messages and traditional mailed letters on increasing participation in research among online patient portal users, as measured by the user joining a research study.

This study tests the hypothesis that at one year follow-up, various user engagement tools (e.g. messaging, banners) will increase the proportion of research profiles created by online patient portal users over profiles created by online patient portal users in the absence of those interventions.

ELIGIBILITY:
Inclusion Criteria:

* Has an account with the online patient portal
* Has logged into the online patient portal at least once in the past year
* Has not set up a research profile

Exclusion Criteria:

* Currently enrolled in a clinical trial
* Opted out of research
* Has received a direct to patient recruitment message within the past year
* On active cancer treatment
* Active member of the study team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 726199 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Number of patients who create a research profile | 12 months
  The outcome will be assessed by querying the patient's electronic medical record to determine whether the patient has registered in the Yale University Volunteer Database. This database is comprised of patients who agree to be contacted if there is a study at Yale that meets their interests.

SECONDARY OUTCOMES:
Number of patients who enroll in a research study | 12 months
  The outcome will be assessed by querying our clinical trials management system or electronic health record system to determine if the patient has consented to participate in a research study.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Smith, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States